CLINICAL TRIAL: NCT05928468
Title: To Evaluate the Safety and Immunogenicity Following a Heterologous Booster Dose of Recombinant SARS-CoV-2 Trivalent Vaccine (CHO Cell) LYB002 in Chinese Adults 18 Years and Above Completed Three-dose Inactivated COVID-19 Vaccine
Brief Title: The Safety and Immunogenicity Following a Heterologous Booster Dose of Recombinant SARS-CoV-2 Vaccine LYB002
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangzhou Patronus Biotech Co., Ltd. (Industry)
Collaborators: Yantai Patronus Biotech Co., Ltd. (Industry); Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LYB002/CT-CHN-IIT02
Record Dates: First submitted 2023-06-29; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LYB002V14 (Experimental): The vaccine LYB002V14 was administered through intramuscular injection.
  Interventions: Biological: LYB002V14
- LYB002V14A (Active Comparator): The vaccine LYB002V14A was administered through intramuscular injection.
  Interventions: Biological: LYB002V14A
- LYB002CA (Active Comparator): The vaccine LYB002CA was administered through intramuscular injection.
  Interventions: Biological: LYB002CA

INTERVENTIONS:
Biological: LYB002V14 — Participants receiving one or two boost doses of LYB002V14 after a three-dose primary series of inactivated COVID-19 vaccine.
  Arms: LYB002V14
Biological: LYB002V14A — Participants receiving one or two boost doses of LYB002V14A after a three-dose primary series of inactivated COVID-19 vaccine.
  Arms: LYB002V14A
Biological: LYB002CA — Participants at 18-59 years old receiving two boost doses of LYB002CA after a three-dose primary series of inactivated COVID-19 vaccine.
  Arms: LYB002CA

SUMMARY:
To evaluate the safety, humoral immunogenicity, cellular immunogenicity and immune persistence following a heterologous booster dose of recombinant SARS-CoV-2 trivalent vaccine (CHO Cell) LYB002 in Chinese adults 18 years and above completed three-dose Inactivated COVID-19 vaccine;

DETAILED DESCRIPTION:
Main Objective

1. To evaluate the safety following a heterologous booster dose of recombinant SARS-CoV-2 trivalent vaccine (CHO Cell) LYB002 in Chinese adults 18 years and above completed three-dose Inactivated COVID-19 vaccine;
2. To evaluate the humoral immunogenicity following a heterologous booster dose of recombinant SARS-CoV-2 trivalent vaccine (CHO Cell) LYB002 in Chinese adults 18 years and above completed three-dose Inactivated COVID-19 vaccine;

Secondary Objectives To evaluate the immune persistence following a heterologous booster dose of recombinant SARS-CoV-2 trivalent vaccine (CHO Cell) LYB002 in Chinese adults 18 years and above completed three-dose Inactivated COVID-19 vaccine;

For exploratory purposes To evaluate the cellular immunogenicity following a heterologous booster dose of recombinant SARS-CoV-2 trivalent vaccine (CHO Cell) LYB002 in Chinese adults 18 years and above completed three-dose Inactivated COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18-59 years, including both males and females;
2. Subjects who agree to participate in this clinical trial voluntarily and sign the informed consent form, are capable of providing valid identification, understanding and complying with the requirements of the clinical protocol.
3. Subjects who have completed three-dose inactivated COVID-19 vaccine at 6 months earlier;
4. S-protein binding antibody IgG concentration was less than 300BAU/mL before booster vaccination in cohort 1, while S-protein binding antibody IgG concentration was not screened in cohort 2; Subjects in cohort 1 and cohort 2 were negative in nucleic acid test or antigen test before booster vaccination.
5. For female participants of childbearing potential, effective contraception measures should be used within 2 weeks prior to participation in this study and the results of pregnancy test is required to be negative. Participants should voluntarily agree to use effective contraceptive measures from the time of signing the informed consent form to the end of the study (effective contraceptive measures including oral contraceptives (excluding emergency contraceptives), injectable or implantable contraceptives, sustained-release topical contraceptives, hormonal patches, intrauterine device, sterilization, abstinence, condoms (for males), diaphragms, cervical caps, etc.).

Exclusion Criteria:

1. Receipt of any COVID-19 prophylactic medication, or previous vaccination history other than other than three doses of inactivated vaccination;
2. Abnormal vital signs with clinical significance prior to enrolment, systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg (systolic blood pressure ≥150mmHg and/or diastolic blood pressure ≥100mmHg for subjects aged ≥60 years), or axillary body temperature ≥37.3℃;
3. The results of laboratory tests before enrollment were abnormal and clinically significant as judged by clinicians;
4. Known allergy, or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients;
5. History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS);
6. Administration of antipyretics, painkillers or anti-allergy drugs within 24 hours prior to enrolment;
7. Receipt of any live attenuated vaccine within 28 days prior to vaccination and other vaccines, such as subunit and inactivated vaccine within 14 days prior to vaccination;
8. Receipt of blood or blood-related products, including immunoglobulins, within 3 months prior to vaccination; or any planned use during the study period.
9. Subjects with the following diseases:

   1. Any acute diseases or acute attacks of chronic diseases within 7 days prior to enrolment；
   2. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.；
   3. Congenital or acquired immunodeficiency or autoimmune disease, or long-term receipt (>14 consecutive days) of glucocorticoid (reference value for dose: ≥20 mg/day prednisone or equivalent) or other immunosuppressive agents within the past 6 months, with exception of inhaled or topical steroids, or short-term use (≤14 consecutive days) of oral corticosteroids；
   4. Currently suffering from or diagnosed with infectious diseases, positive screening results for hepatitis B surface antigen, hepatitis C antibody, treponema pallidum antibody, human immunodeficiency virus antibody；
   5. History or family history of neurological disorders (convulsions, epilepsy, encephalopathy, etc.) or psychiatric disorders；
   6. Asplenia, or functional asplenia；
   7. Presence of severe, uncontrollable or hospitalized cardiovascular diseases, diabetes, blood and lymphatic diseases, immune diseases, liver and kidney diseases, respiratory diseases, metabolic and skeletal diseases, or malignant tumors;
   8. Contraindications to IM injections and blood draws, such as coagulation disorders, thrombotic or bleeding disorders, or conditions that needs continuous anticoagulant usage.
10. Drug or alcohol abuse (alcohol intake ≥ 14 units per week) which in the investigator's opinion would compromise the participant's safety or compliance with the study procedures;
11. Pregnant or lactating females;
12. Having participated or participating in COVID-19 related clinical trials, and those participating or planning to participate in other clinical trials during the study period;
13. Presence of any underlying disease or condition which, in the opinion of the investigator, may place the subject at unacceptable risk, is unable to meet the requirements of the protocol, or interfere with the assessment of vaccine response.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
The frequencies and percentages of adverse events within 30 minutes of each booster dose | within 30 minutes after booster vaccination
  Statistical description of solicited and unsolicited adverse events (AEs) will be listed.Frequencies and percentages of AEs, including overall AEs, AEs related tovaccination, AEs classified as grade 3 or worse, AEs classified as grade 3 or worsethat related to vaccination, AEs leading to participant's withdrawal, AEs leading toparticipant's withdrawal that related to vaccination will be presented. Fisher's exacttest will be used to compare the differences between the groups.
  Solicited and unsolicited AEs within 30 mins after vaccination will be collected
The frequencies and percentages of adverse events within 7 days of each booster dose | 7 days after booster vaccination
  Statistical description of solicited and unsolicited adverse events (AEs) will be listed.Frequencies and percentages of AEs, including overall AEs, AEs related tovaccination, AEs classified as grade 3 or worse, AEs classified as grade 3 or worsethat related to vaccination, AEs leading to participant's withdrawal, AEs leading toparticipant's withdrawal that related to vaccination will be presented. Fisher's exacttest will be used to compare the differences between the groups.
  Solicited local/systemic AEs within 7 days of booster dose will be collected
The frequencies and percentages of adverse events within 28 days of each booster dose | 28 days after booster vaccination
  Statistical description of solicited and unsolicited adverse events (AEs) will be listed.Frequencies and percentages of AEs, including overall AEs, AEs related tovaccination, AEs classified as grade 3 or worse, AEs classified as grade 3 or worsethat related to vaccination, AEs leading to participant's withdrawal, AEs leading toparticipant's withdrawal that related to vaccination will be presented. Fisher's exacttest will be used to compare the differences between the groups.
  Unsolicited AEs within 28 days of booster dose will be collected
The Seroconversion (SCRs) of neutralizing antibodies (Nabs) and S protein-bindingantibodies at 14 days after each booster immunization | 14 days after each booster vaccination
  The Seroconversion (SCRs) with Clopper-Pearson 95% CIs of neutralizing antibodies(Nabs) against prototype SARS-CoV-2 and circulating VOCs using Vesicularstomatitis virus (VSV)-based pseudovirus neutralizing assays, S protein-bindingantibodies using ELISA assays, at 14 days after each booster immunization will be calculated for each group, compared with the baseline.
The Seroconversion (SCRs) of neutralizing antibodies (Nabs) and S protein-bindingantibodies at 28 days after each booster immunization | 28 days after each booster vaccination
  The Seroconversion (SCRs) with Clopper-Pearson 95% CIs of neutralizing antibodies(Nabs) against prototype SARS-CoV-2 and circulating VOCs using Vesicularstomatitis virus (VSV)-based pseudovirus neutralizing assays, S protein-bindingantibodies using ELISA assays, at 28 days after each booster immunization will be calculated for each group, compared with the baseline.
The Geometric Neutralizing titers (GMT) of neutralizing antibodies (Nabs) and Sprotein-binding antibodies at 14 days after each booster vaccination | 14 days after each booster vaccination
  The Geometric Neutralizing titers (GMT) with Clopper-Pearson 95% CIs ofneutralizing antibodies (Nabs) against prototype SARS-CoV-2 and circulating VOCsusing Vesicular stomatitis virus (VSV)-based pseudovirus neutralizing assays, Sprotein-binding antibodies using ELISA assays, at baseline, at 14 days after the booster immunization will be calculated for each group, compared with the baseline.
The Geometric Neutralizing titers (GMT) of neutralizing antibodies (Nabs) and Sprotein-binding antibodies at 28 days after each booster vaccination | 28 days after each booster vaccination
  The Geometric Neutralizing titers (GMT) with Clopper-Pearson 95% CIs ofneutralizing antibodies (Nabs) against prototype SARS-CoV-2 and circulating VOCsusing Vesicular stomatitis virus (VSV)-based pseudovirus neutralizing assays, Sprotein-binding antibodies using ELISA assays, at baseline, at 28 days after the booster immunization will be calculated for each group, compared with the baseline.
The Geometric mean fold rise (GMFR) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 14 days after the booster immunization | 14 days after each booster vaccination
  The Geometric mean fold rise (GMFR) with Clopper-Pearson 95% CIs of neutralizingantibodies (Nabs) against prototype SARS-CoV-2 and circulating VOCs usingVesicular stomatitis virus (VSV)-based pseudovirus neutralizing assays, S protein-binding antibodies using ELISA assays, at baseline, at 14 days after the booster immunization will be calculated for each group, compared with the baseline.
The Geometric mean fold rise (GMFR) of neutralizing antibodies (Nabs) and S protein-binding antibodies at 28 days after the booster immunization | 28 days after each booster vaccination
  The Geometric mean fold rise (GMFR) with Clopper-Pearson 95% CIs of neutralizingantibodies (Nabs) against prototype SARS-CoV-2 and circulating VOCs usingVesicular stomatitis virus (VSV)-based pseudovirus neutralizing assays, S protein-binding antibodies using ELISA assays, at baseline, at 28 days after the booster immunization will be calculated for each group, compared with the baseline.

SECONDARY OUTCOMES:
The Seroconversion (SCRs) of neutralizing antibodies (Nabs) and S protein-binding | 3 months after the last booster vaccination
  The Seroconversion (SCRs) with Clopper-Pearson 95% CIs of neutralizing antibodies(Nabs) against prototype SARS-CoV-2 and circulating VOCs using Vesicularstomatitis virus (VSV)-based pseudovirus neutralizing assays, S protein-bindingantibodies using ELISA assays, at 3 months after the last booster immunization will be calculated for all participants.
The Geometric Neutralizing titers (GMT) of neutralizing antibodies (Nabs) and GMC of Sprotein-binding antibodies | 3 months after the last booster vaccination
  The Geometric Neutralizing titers (GMT) with Clopper-Pearson 95% CIs ofneutralizing antibodies (Nabs) against prototype SARS-CoV-2 and circulating VOCsusing Vesicular stomatitis virus (VSV)-based pseudovirus neutralizing assays, the GMC of Sprotein-binding antibodies using ELISA assays, at 3 months after the last booster immunization will be calculated for all participants.
The Geometric mean fold rise (GMFR) of neutralizing antibodies (Nabs) and S protein-binding antibodies | 3 months after the last booster vaccination
  The Geometric mean fold rise (GMFR) with Clopper-Pearson 95% CIs of neutralizingantibodies (Nabs) against prototype SARS-CoV-2 and circulating VOCs usingVesicular stomatitis virus (VSV)-based pseudovirus neutralizing assays, S protein-binding antibodies using ELISA assays, at 3 months after the last booster immunization will be calculated for all participants.
The frequencies and percentages of adverse events | 6 months after the last booster vaccination
  The incidence of serious adverse events (SAE) and adverse events of special interest (AESI) in all participants within 6 months after the last booster dose;
The changes of the frequencies and percentages of adverse events from the baseline at the 3rd day after each boost vaccination | 3 days after each booster vaccination
  the changes of laboratory tests on the third day after each dose of booster vaccination compared with those before vaccination

OTHER OUTCOMES:
The counts of spot forming cells (SFCs) per 3×105 peripheral blood mononuclear cells(PBMCs) of Cellular immunity | 14 days after each booster vaccination
  RBD-specific IFN-γ, IL-2, and IL-4 cytokine levels before and 14 days after each dose of booster vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolan Yong, Bachelor, Principal Investigator — Affiliated Hospital to North Sichuan MedicalCollege
Locations (1):
- Affiliated Hospital of North Sichuan MedicalCollege, Chengdu, Sichuan, China